CLINICAL TRIAL: NCT01999244
Title: Impact of Self-Monitoring Technology and Interventionist Contact on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 209313; F32DK100069-01 (NIH)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Weight Loss; Self-monitoring; Food Records; Self-weighing; Technology
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Technology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SC (Experimental): Self-guided self-monitoring condition. Participants will receive standard self-monitoring tools and information on weight regulation.
  Interventions: Behavioral: Self-monitoring skills
- TECH (Experimental): Technology condition. Participants will receive self-monitoring technology and information regarding weight regulation.
  Interventions: Behavioral: Self-monitoring skills; Behavioral: Technology
- TECH+INT (Experimental): Technology plus interventionist contact arm. Participants will receive self-monitoring technology, information regarding weight regulation, and interventionist contact via telephone.
  Interventions: Behavioral: Self-monitoring skills; Behavioral: Technology; Behavioral: Interventionist Contact

INTERVENTIONS:
Behavioral: Self-monitoring skills
Behavioral: Technology
  Arms: TECH; TECH+INT
Behavioral: Interventionist Contact
  Arms: TECH+INT

SUMMARY:
Despite continued research on effective interventions, obesity remains a major public health issue in the United States. Current treatments, including behavioral weight management programs, weight loss surgery, and pharmacotherapy, tend to be high in cost and have limited reach, reducing the ability of these treatments to address the population-wide scope of the obesity epidemic. Recent advances in technology that improve the ease of self-monitoring and provide targeted feedback offer promise to help larger groups of individuals to lose weight. Despite the commercial popularity of these products, however, little research has been conducted to evaluate their impact on excess body weight or to determine how they should ideally be implemented. Two key questions need to be addressed. First, is use of self-monitoring technology sufficient to produce weight loss, or must this technology be combined with interventionist contact? Second, how cost-effective is a technology-based intervention, with and without interventionist contact? The current study is small prospective, randomized pilot study comparing a self-guided self-monitoring condition (SC) to a technology only condition (TECH) and a technology plus interventionist support condition (TECH+INT). All participants will all be given basic weight management information knowledge and randomized to one of three conditions. Participants in the self-guided self-monitoring condition (SC) will receive traditional paper self-monitoring logs, a standard body weight scale, and a pedometer and calorie book; participants in the technology-based condition (TECH) will receive an electronic activity monitor and WiFi-enabled body weight scale, and will track caloric intake via an associated website; and participants in the interventionist contact condition (TECH+INT) will receive the same technology as in the TECH condition, combined with weekly interventionist contact delivered via telephone. We will compare the impact of each condition on weight loss and investigate preliminary cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* BMI between 27 and 40 kg/m2
* Access to a computer and WIFI in the home

Exclusion Criteria:

* Weight over 340 lbs
* Physical limitations that prevent walking 1/4 mile without stopping
* Currently participating in another weight loss program or taking weight loss medication
* Currently pregnant, lactating, less than 6-months post-partum, or plans to become pregnant during the 6-month study period
* Uncontrolled hypertension or diabetes
* History of coronary heart disease
* Terminal Illness
* Plans to relocate during the 6-month study period
* Substance Abuse
* Severe psychiatric disorders
* Dementia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Weight | 6 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Ross, PhD MPH, Principal Investigator — The Miriam Hospital; Rena R Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control & Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Chhabria K, Ross KM, Sacco SJ, Leahey TM. The Assessment of Supportive Accountability in Adults Seeking Obesity Treatment: Psychometric Validation Study. J Med Internet Res. 2020 Jul 28;22(7):e17967. doi: 10.2196/17967. PMID 32720911
- [Derived] Ross KM, Wing RR. Impact of newer self-monitoring technology and brief phone-based intervention on weight loss: A randomized pilot study. Obesity (Silver Spring). 2016 Aug;24(8):1653-9. doi: 10.1002/oby.21536. Epub 2016 Jul 1. PMID 27367614